CLINICAL TRIAL: NCT02286674
Title: Use of Handheld Audiovisual Devices to Treat Pediatric Preoperative Anxiety: A Randomized Control Trial.
Brief Title: Use of Handheld Audiovisual Devices to Treat Pediatric Preoperative Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McLaren Health Care (Other)
Responsible Party: Principal Investigator, MCRI Staff, Michael Stein, McLaren Health Care
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201400076
Record Dates: First submitted 2014-10-10; First posted 2014-11-10 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Pediatric Preoperative Anxiety
Keywords: mYpas; anxiety; distraction; inhalation induction
MeSH Terms: conditions — Anxiety Disorders | interventions — Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tablet for watching movie (Experimental): The study group will receive standard of care in addition to a tablet to watch movies and/or TV
  Interventions: Other: Tablet (Audio/Visual Device)
- Standard of care - no tablet (No Intervention): The control group will receive standard of care only.

INTERVENTIONS:
Other: Tablet (Audio/Visual Device) — Subjects will be given a tablet to use before surgery
  Arms: Tablet for watching movie

SUMMARY:
Anxiety in children undergoing surgery is a central concern to both parents and healthcare workers, including nurses, surgeons, and anesthesiologists. It has been ranked by anesthesiologists as one of the top five important low-morbidity anesthesia outcomes (1). This study would determine whether such devices would decrease anxiety in children prior to induction of anesthesia for outpatient surgery. Two hundred children ages 2-12 will be enrolled.

DETAILED DESCRIPTION:
Anxiety in children undergoing surgery is a central concern to both parents and healthcare workers, including nurses, surgeons, and anesthesiologists. It has been ranked by anesthesiologists as one of the top five important low-morbidity anesthesia outcomes (1). Extensive research has been done characterizing, quantifying, and risk stratifying anxiety in this group as well as identifying a multitude of treatment options both pharmacological and nonpharmacological. Up to 60% of all children develop anxiety in the preoperative holding area and during anesthetic induction (2). The incidence can be much higher in some subpopulations. Preoperative anxiety has been attributed to number of causes including separation from parents and uncertainty about anesthesia, the procedure, and outcome (3).

Interestingly, anxiety prior to surgery has effects that extend into the intraoperative, acute recovery and subacute recovery timeframes. Patients with high levels of preoperative anxiety have been found to require greater anesthetic dosages (4). There is a higher incidence of emergence delirium in children with higher levels of preoperative anxiety (5, 6). These patients also have with a higher incidence of postoperative pain and require more analgesic medications (7). Furthermore, there are well documented maladaptive behavioral changes that can occur in 30-54% of children two weeks following surgery (8). These include generalized anxiety, nighttime crying, enuresis, separation anxiety, and temper tantrums. Twenty percent of these children maintain this behavior at 6 months and 7% persist at 1 year after the operation (9). High preoperative anxiety levels correlate with these behavior changes (2, 5, 8,10).

Many other interventions have been tried to decrease anxiety with varying success. Most are aimed at distraction. Music therapy appears to be therapist-dependent (12). Hand held video games appear to help decrease anxiety, even during induction (13). Even having clowns in the operating room at induction of anesthesia seems to help -- the study concluded that staff were quite resistant to maintaining the clown program (14). Interestingly, a small randomized controlled trial showed that parents distracting their children during induction with novel toys and books or blowing bubbles did not decrease anxiety (15).

Few studies have considered the use of tablets as distraction tools for children undergoing surgery. Low and Pittaway briefly described using an iPhone™ to distract 93 children in the preoperative period (16). However, the results are simply anecdotal. Patel et al. described a randomized control trial using hand held video games as a means of distraction compared to midazolam and a control group. They used the well validated and extensively used modified Yale Preoperative Anxiety Score (17) to measure anxiety levels. However, this study included parents being present at induction in all the groups, which may make the results difficult to apply at the majority of institutions, where parental presence is not used - our institution included (11).

In addition, premedication may be given to 50% of patients nationally, but it is not popular among parents (11,18). If the majority of practitioners do not use parental presence at induction, preoperative education programs are not yet in widespread use and half of patients are not premedicated, that leaves a significant portion of the population with little intervention for the time of separation and for time of induction of anesthesia. Finding an economical, efficient means to help decrease anxiety without high doses of premedication would be quite appealing.

This study would determine whether such devices would decrease anxiety in children prior to induction of anesthesia for outpatient surgery. Two hundred children ages 2-12 will be enrolled. Half would be in the control group, which would receive standard care. Half would be in the study group, which would receive a tablet device in the preoperative holding area and would be allowed to watch TV or movies from a preloaded list until they are given anesthetic gases in the operating room. The subjects would be observed for outward signs of anxiety and scored using a well validated and well used anxiety scale, the modified Yale preoperative anxiety scale, at several points in time prior to induction of anesthesia. The expected total study length is 6 months based on the current number of pediatric cases at the study site.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 2-12
2. Outpatient surgery procedures
3. ASA I of II (No or mild systemic disease)
4. Parental/guardian ability to understand and willingness to sign written informed consent
5. Patient assent to use tablet, if they are randomized to the study group
6. Anesthetic plan includes sevoflurane inhalation induction as determined by the anesthesiologist

Exclusion Criteria:

1. Psychoactive medications (e.g. antipsychotics, mood stabilizers, anxiolytics, antidepressants, narcotics)
2. Diagnosed psychiatric disease
3. Developmental disabilities
4. History of photosensitive seizures
5. Patient requiring sedative or narcotic medications prior to induction of anesthesia, as determined by the anesthesiologist.
6. Parental/guardian inability to understand or refusal to sign written informed consent
7. Patient unwillingness or inability to use tablet
8. Anesthetic plan does not include sevoflurane induction, as determined by anesthesiologist.
9. Non English speaking patient and/or parent/guardian

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2014-11; Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Yale Preoperative Anxiety Score | Baseline
  Anytime prior to patient being ifnormed of group assignment
Yale Preoperative Anxiety Score | Upon patient spearation from parents Approx 15-20 minutes
  Approx 15-20 minutes after the study group participants receive a tablet
Yale Preoperative Anxiety Score | Patient enters operating room 1-32 minutes
  1-32 minutes after #2
Yale Preoperative Aniety Score | Placement of face mask on patient ofr anesthetic delivery 1-2 minutes
  1-2 minutes after #3

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stein, DO, Principal Investigator — Physician
Locations (1):
- McLaren Greater Lansing Hospital, Lansing, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Macario A, Weinger M, Truong P, Lee M. Which clinical anesthesia outcomes are both common and important to avoid? The perspective of a panel of expert anesthesiologists. Anesth Analg. 1999 May;88(5):1085-91. doi: 10.1097/00000539-199905000-00023. PMID 10320175
- [Background] Kain ZN, Mayes LC, O'Connor TZ, Cicchetti DV. Preoperative anxiety in children. Predictors and outcomes. Arch Pediatr Adolesc Med. 1996 Dec;150(12):1238-45. doi: 10.1001/archpedi.1996.02170370016002. PMID 8953995
- [Background] Kain ZN, Caldwell-Andrews A, Wang SM. Psychological preparation of the parent and pediatric surgical patient. Anesthesiol Clin North Am. 2002 Mar;20(1):29-44. doi: 10.1016/s0889-8537(03)00053-1. PMID 11892508
- [Background] Maranets I, Kain ZN. Preoperative anxiety and intraoperative anesthetic requirements. Anesth Analg. 1999 Dec;89(6):1346-51. doi: 10.1097/00000539-199912000-00003. PMID 10589606
- [Background] Kain ZN, Caldwell-Andrews AA, Maranets I, McClain B, Gaal D, Mayes LC, Feng R, Zhang H. Preoperative anxiety and emergence delirium and postoperative maladaptive behaviors. Anesth Analg. 2004 Dec;99(6):1648-1654. doi: 10.1213/01.ANE.0000136471.36680.97. PMID 15562048
- [Background] Aono J, Mamiya K, Manabe M. Preoperative anxiety is associated with a high incidence of problematic behavior on emergence after halothane anesthesia in boys. Acta Anaesthesiol Scand. 1999 May;43(5):542-4. doi: 10.1034/j.1399-6576.1999.430509.x. PMID 10342002
- [Background] Kain ZN, Mayes LC, Caldwell-Andrews AA, Karas DE, McClain BC. Preoperative anxiety, postoperative pain, and behavioral recovery in young children undergoing surgery. Pediatrics. 2006 Aug;118(2):651-8. doi: 10.1542/peds.2005-2920. PMID 16882820
- [Background] Kain ZN, Wang SM, Mayes LC, Caramico LA, Hofstadter MB. Distress during the induction of anesthesia and postoperative behavioral outcomes. Anesth Analg. 1999 May;88(5):1042-7. doi: 10.1097/00000539-199905000-00013. PMID 10320165
- [Background] Kain ZN, Mayes LC, Wang SM, Hofstadter MB. Postoperative behavioral outcomes in children: effects of sedative premedication. Anesthesiology. 1999 Mar;90(3):758-65. doi: 10.1097/00000542-199903000-00018. PMID 10078677
- [Background] Karling M, Stenlund H, Hagglof B. Child behaviour after anaesthesia: associated risk factors. Acta Paediatr. 2007 May;96(5):740-7. doi: 10.1111/j.1651-2227.2007.00258.x. PMID 17462064
- [Background] Kain ZN, Caldwell-Andrews AA, Krivutza DM, Weinberg ME, Wang SM, Gaal D. Trends in the practice of parental presence during induction of anesthesia and the use of preoperative sedative premedication in the United States, 1995-2002: results of a follow-up national survey. Anesth Analg. 2004 May;98(5):1252-9, table of contents. doi: 10.1213/01.ane.0000111183.38618.d8. PMID 15105196
- [Background] Kain ZN, Caldwell-Andrews AA, Krivutza DM, Weinberg ME, Gaal D, Wang SM, Mayes LC. Interactive music therapy as a treatment for preoperative anxiety in children: a randomized controlled trial. Anesth Analg. 2004 May;98(5):1260-6, table of contents. doi: 10.1213/01.ane.0000111205.82346.c1. PMID 15105197
- [Background] Patel A, Schieble T, Davidson M, Tran MC, Schoenberg C, Delphin E, Bennett H. Distraction with a hand-held video game reduces pediatric preoperative anxiety. Paediatr Anaesth. 2006 Oct;16(10):1019-27. doi: 10.1111/j.1460-9592.2006.01914.x. PMID 16972829
- [Background] Vagnoli L, Caprilli S, Robiglio A, Messeri A. Clown doctors as a treatment for preoperative anxiety in children: a randomized, prospective study. Pediatrics. 2005 Oct;116(4):e563-7. doi: 10.1542/peds.2005-0466. PMID 16199685
- [Background] Watson A, Srinivas J, Daniels L, Visram A. Preparation of parents by teaching of distraction techniques does not reduce child anxiety at anaesthetic induction. Paediatr Anaesth 2002;12:823-824.
- [Background] Low DK, Pittaway AP. The 'iPhone' induction - a novel use for the Apple iPhone. Paediatr Anaesth. 2008 Jun;18(6):573-4. doi: 10.1111/j.1460-9592.2008.02498.x. Epub 2008 Feb 28. No abstract available. PMID 18312515
- [Background] Kain ZN, Mayes LC, Cicchetti DV, Bagnall AL, Finley JD, Hofstadter MB. The Yale Preoperative Anxiety Scale: how does it compare with a "gold standard"? Anesth Analg. 1997 Oct;85(4):783-8. doi: 10.1097/00000539-199710000-00012. PMID 9322455
- [Background] Kain ZN, Caldwell-Andrews AA, Wang SM, Krivutza DM, Weinberg ME, Mayes LC. Parental intervention choices for children undergoing repeated surgeries. Anesth Analg. 2003 Apr;96(4):970-975. doi: 10.1213/01.ANE.0000055650.54661.12. PMID 12651644